CLINICAL TRIAL: NCT04815616
Title: Efficacy of Capecitabine With Adjuvant Radiotherapy in Treatment of Early Stages Breast Cancer (Retrospective Study).
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Adel Ali, Principal investigator, Assiut University
Other Study IDs: Radiotherapy in breast cancer
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Radiotherapy — Capecitabine with adjuvant radiotherapy in treatment of Early Stages Breast Cancer

SUMMARY:
1- Determine the efficacy and safety of concurrent capecitabine and external beam irradiation in patients with early stages breast cancer.

DETAILED DESCRIPTION:
Breast cancer is the most commonly diagnosed cancer among American women, In 2021 it is estimated that about 30%of newly diagnosed cancers in women will be breast cancer. As of January 2021, there are more than 3,8 million women with history of breast cancer in U.S.A including women currently being treated and those who finished treatment.

Death rates have been steady in women under 50years old since 2007,but have continued to drop in women over 50 years old .The overall death rate from breast cancer decreased by 1% per year from 2013 to 2018.these decreases are thought to be the result of treatment advances and earlier detection and screening.

About 43,600 women in U.S.A are expected to die in 2021 from Breast cancer. A woman's risk of breast cancer nearly doubles if she has a first degree relative who has been diagnosed with breast cancer .Less than 15% of women who get breast cancer have family member diagnosed with breast cancer. About 85% of breast cancer occur in women who have no family history of breast cancer ,these occurs due to genetic mutations that happen as results of aging process rather than inherited mutations. . [1]

The treatment of breast cancer includes the treatment of local disease with surgery, radiation therapy or both ,and systemic treatment with chemotherapy ,endocrine therapy ,biologic therapy or combination of these.[2]

After lumpectomy, whole breast irradiation is strongly recommended with or without boost to tumor bed for node positive (category 1 for those with positive nodes; category 2A for those with negative axillary nodes). This recommendation shows reduction in 10 -year risk of recurrence in those who received whole breast irradiation versus those who did not. In addition significant reduction in 15-year risk of breast cancer death was also observed. [3] Radiotherapy after mastectomy and Axillary lymph node dissection in (node positive disease) reduced both recurrence and breast cancer mortality in women with 1-3 positive lymph nodes even when systemic therapy was administered. [4] In node negative disease and tumor less than 5 cm and clear margin >1mm, post mastectomy radiation therapy is not recommended.

Primary radiotherapy has been used for local control of breast tumors in variety of situations. Excellent local control was obtained by Chargari et al with radiation alone in early stage tumors with loco regional control at 7 years of 95,8%. [5] Certain chemotherapeutic agents are known as radio-sensitizers, allowing for enhanced therapeutic ratio and improved tumor control when given concurrently with radiotherapy .concurrent chemo -radiotherapy has been used at multiple disease sites , with gains in local control, disease free survival ,and overall survival over radiation alone.[6] Combining adjuvant radiotherapy with capecitabine appears to be safe and feasible for chemotherapy resistant breast cancer patient with stage I-III who has residual disease in form of improve local and distant disease control [7].

ELIGIBILITY:
Inclusion Criteria:

1. Age of patients ≥ 18 years old patients.
2. Histopathology confirmed: invasive ductal carcinoma.
3. Breast conservative surgery or mastectomy.
4. Early stage breast cancer patients.
5. Adjuvant chemotherapy in the form of Anthracyclins based.

Exclusion Criteria:

1. Contraindications to radiotherapy: such as previous irradiation to chest wall or skin diseases.
2. Pregnancy or lactation.
3. Contraindications to capecitabine such as: severe renal impairment Or hypersensitivity to capecitabine.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early stage breast cancer Patients who received adjuvant Radiotherapy with capecitabine .
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | baseline
  Disease free survival

REFERENCES:
- [Background] 1-. American Cancer society. .American cancer society. Cancer facts and figures 2021.available at: How common is breast cancer/ Jan 2021. http://www.cancer.org/content/dam/cancer-org/research/cancer-fact and ststics /annual- cancer-facts-and figures -2021.pdf. 2- stackievicz R ,Paran H ,Bernhiem J, et al. Prognostic significance of HER-2 /neu expression in patients with ductal carcinoma in situ. Isr med assoc j 2010 ;12:290-295 available at : http://www.ncbi.nlm.nih.gov,pubmed/20929083. 3-. early breast cancer trialists collaborative G, Darby S,Mc Gale P,et al. effect of radiotherapy after breast conserving surgery on 10-year recurrence and 15- year breast cancer death :meta-analysis of individual patients data for 10,801 women in 17 randomized trials .Lancet 2011;378:1707-1716 Available at: http:// www.ncbi.nlm.nih.gov,pubmed/22019144. 4-.early breast cancer trialists collaborative G, Darby S,Mc Gale P,et al. effect of radiotherapy after mastectomy and axillary surgery on 10- year recurrence and 20-year breast cancer mortality :meta-analysis individual patients data for 8135 women in 22 randomized trials. Lancet 2014; 383:2127-2135 available at: http:// www.ncbi.nlm.nih.gov,pubmed/24656685. 5-.Chargari C,Kirova YM,Laki F, et al. the impact of loco regional treatment in elderly breast cancer patients :hypo -fractionated exclusive radiotherapy, single institution long term results .breast 2010 ;19;413-6. 6-.Karasawa K,Saito M, Hariwatari H et al. the role of chemo radiotherapy in patients with unresectable T4 breast tumors breast cancer 2013;20:254-61. 7- N Engl J Med 2017; 376:2147-2159